CLINICAL TRIAL: NCT01634802
Title: Evaluation of Use of Clinical Decision Support System for Early Detection of Immunological Treatment Failure Among HIV Patients in Resource Constrained Settings
Brief Title: Evaluation of Use of Clinical Decision Support System in HIV Care in Resource Constrained Settings
Acronym: CDSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Tom Oluoch, Mr., Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2073
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: HIV
Keywords: Clinical Decision Support Systems; Electronic Medical Record; Resource constrained countries; HIV
MeSH Terms: interventions — Electronic Health Records

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMR Only (No Intervention): Clinics in this arm of the study will have a standard Electronic Medical Record (EMR) system installed - without a computerized decision support system.
  Interventions: Other: EMR Only
- EMR+CDSS (Experimental): Clinics in this arm of the study will have an Electronic Medical Record (EMR) system with Clinical Decision Support System (CDSS) enhancement implemented as alerts to aid the clinician in decision making.
  Interventions: Other: EMR+CDSS

INTERVENTIONS:
Other: EMR Only — Clinics in this arm of the study will have a standard Electronic Medical Record (EMR) system installed - without a computerized decision support system.
  Arms: EMR Only
Other: EMR+CDSS — Clinics in this arm of the study will have an Electronic Medical Record (EMR) system with Clinical Decision Support System (CDSS) enhancement implemented as alerts to aid the clinician in decision making.
  Other Names: Clinical Decision Support Systems; Electronic Medical Records
  Arms: EMR+CDSS

SUMMARY:
The purpose of this study is to determine whether the use of a Computerized Decision Support System (CDSS) in form of alerts to clinicians enhances early detection of immunological treatment failure in HIV patients.

DETAILED DESCRIPTION:
We hypothesize that there is no difference in the time to detecting immunological treatment failure among HIV patients in resource poor settings whether the clinicians use an Electronic Medical Record (EMR) system with a Computerized Decision Support (CDSS) or an EMR without a CDSS. In this study, 20 clinics were assigned to the intervention (EMR+CDSS) arm and non-intervention arm (EMR only) and will be followed up for 12 months to assess whether there are any differences in time taken to detect immunological treatment failure based on CD4 cell count.

ELIGIBILITY:
Inclusion Criteria:

* All HIV patients enrolled in participating clinics

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1460 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The main end-point of the study will be the proportion of patients on treatment who have experienced treatment failure and appropriate clinical action taken according to the guidelines. | 12 months

SECONDARY OUTCOMES:
Other outcome measures will be the proportion of CD4 cell counts done on time and proportion of pre-ART patient eligible for treatment that are initiated within 30 days of eligibility. The median time taken to clinical action will be measured. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Oluoch, MSc, Principal Investigator — Centers for Disease Control and Prevention; Daniel Kwaro, MD, Principal Investigator — KEMRI-CDC
Locations (1):
- KEMRI/CDC Clinical Research Center, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Oluoch T, Cornet R, Muthusi J, Katana A, Kimanga D, Kwaro D, Okeyo N, Abu-Hanna A, de Keizer N. A clinical decision support system is associated with reduced loss to follow-up among patients receiving HIV treatment in Kenya: a cluster randomized trial. BMC Med Inform Decis Mak. 2021 Dec 20;21(1):357. doi: 10.1186/s12911-021-01718-0. PMID 34930228
- [Derived] Oluoch T, Katana A, Kwaro D, Santas X, Langat P, Mwalili S, Muthusi K, Okeyo N, Ojwang JK, Cornet R, Abu-Hanna A, de Keizer N. Effect of a clinical decision support system on early action on immunological treatment failure in patients with HIV in Kenya: a cluster randomised controlled trial. Lancet HIV. 2016 Feb;3(2):e76-84. doi: 10.1016/S2352-3018(15)00242-8. Epub 2015 Dec 17. PMID 26847229